CLINICAL TRIAL: NCT01739868
Title: Screening and Understanding of the Pre-diabetes: DECODIAB
Acronym: DECODIAB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 09/9-A
Record Dates: First submitted 2012-11-23; First posted 2012-12-04 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Pre-diabetes
Keywords: Pre-diabetes; Type 2 diabetes; Biomarkers; Diabetes risk score
MeSH Terms: conditions — Glucose Intolerance; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Biopsies of muscular and fat tissue — 3 half days of metabolic exploration including blood sample, urinary taking, OGTT (oral glucose tolerance test), biopsies of muscular and fat tissue:
  * 1 visit the first year (inclusion visit)
  * 1 visit at the end of 5 years of follow-up or in the appearance of type 2 diabetes
  * 1 intermediary visit (in 3 years) or activated by the following conditions:
    * Escalation of the glycemia (increase of 0.1g / l of the glycemia and/or 0.3 % of the HbA1c)
    * Normalization of the glycemia (fasting blood glucose < 1 g/l)

SUMMARY:
The main objective of the study is to understand the pathophysiological mechanisms involved in switching from pre-diabetes to type 2 diabetes and to identify new biomarkers of type 2 diabetes risk in the population of patients with pre-diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years)
* Subjects with diabetes risk score ≥ 12 or with impaired fasting glucose: blood glucose ≥ 1.10 g/l and < 1 .26 g/L
* And with impaired fasting glucose : blood glucose ≥ 1.10 g/l and < 1 .26 g/L ; or blood glucose ≥ 1g/l and < 1,1 g/L WITH HbA1C ≥ 6,5%
* Signed informed consent
* Subjects affiliated with an appropriate social security system

Exclusion Criteria:

* Fasting glycemia ≥ 1.26 g/l
* Fasting glycemia ≤ 1.10 g/l AND HbA1C < 6,5%
* Fasting glycemia < 1 g/l
* Subjects previously treated with oral anti-diabetic: metformin, glitazones, inhibitors of α-glucosidase, sulfonylurea, repaglinide, inhibitors of DPP-IV.
* Subjects previously treated with insulin, except gestational diabetes
* Severe coagulation disorders
* Thrombocytopenia < 100 000/mm 3
* Severe psychiatric disorders
* Severe renal insufficiency (creatinine clearance < 30 ml/min)
* Severe hepatic insufficiency
* Alcohol abuse (> 30g/j)
* Contra-indication in the realization of the local anesthetic
* Subject unable to follow the study during the 5 years of follow-up
* Subject exclusion period in a previous study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2011-04; Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
To identify new biomarkers | 5 years
  The main objective of the study is to understand the pathophysiological mechanisms involved in switching from pre-diabetes to type 2 diabetes and to identify new biomarkers of type 2 diabetes risk in the population of patients with pre-diabetes

SECONDARY OUTCOMES:
To identify new therapeutic targets | 5 years
  To identify new therapeutic targets for the prevention of the appearance of the diabetes in the population of patients with pre-diabetes
To connect identified biomarkers with the degree of insulinoresistance | 5 years
  To connect identified biomarkers with the degree of insulinoresistance (HOMA-R) and with β pancreatic function (IOG) in the population of patients with pre-diabetes.
Number of patients with high Diabetes Risk Score and pre-diabetes | 5 years
  To evaluate the interest of the Diabetes Risk Score in identifying subjects with pre-diabetes in the French population
Number of patients with others cardiovascular risk factors | 5 years
  To evaluate the prevalence of others cardiovascular risk factors associated with pre-diabetes: dyslipidemia, hypertension, metabolic liver disease

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand CARIOU, Pr, Principal Investigator — Nantes University Hospital
Locations (1):
- Nantes University Hospital, Nantes, France